CLINICAL TRIAL: NCT05332769
Title: Cumulus Cell Mitochondrial Activity as a Non-invasive Marker of Embryo Quality
Brief Title: Cumulus Cell Mitochondrial Activity as a Non-invasive Marker of Embryo Quality (FLIM)
Status: Active, not recruiting | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: The Needleman Lab, Northwest Lab Building 359,52 Oxford Street Cambridge MA 02138. (Unknown); Harvard University Faculty of Medicine (Other); Hospital Foch, Suresnes, France. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 11/21/DD/BVMD
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: IVF/ICSI; Frozen Embryo Transfer; Cumulus Cell; Fluorescence Lifetime Imaging Microscopy
Keywords: Cumulus cell; Day 5/6 frozen embryo; Fluorescence lifetime imaging microscopy; FLIM; IVF/ICSI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cumulus cell of oocyte
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile women have IVF/ICSI cycle: All Vietnamese infertile women who have IVF/ICSI cycle with at least 8 follicles ≥ 10 mm on ultrasonography at induced ovulation date agreed to freeze-all day 5-6 embryos at IVFMD and IVFMD PN will be enrolled in the study.
  Interventions: Genetic: FLIM parameters

INTERVENTIONS:
Genetic: FLIM parameters — Cumulus samples (CCs) will be collected following the protocol on the day of oocyte pick up (OPU). CCs are frozen by the cryo-tech method, then stored in liquid nitrogen at -196oC. Information of CC samples and processed date/time is recorded. After all, samples are collected, they will be transferred to The Needleman Lab, Northwest Lab Building 359,52 Oxford Street Cambridge MA 02138 to measure mitochondria metabolism using FLIM.
  Other Names: fluorescence lifetime imaging microscopy

SUMMARY:
This study aims to test the extent of association of FLIM parameters of cumulus cells with clinical outcomes (clinical pregnancy, ongoing pregnancy at 12 weeks, and live birth) of the embryos that result from the enclosed oocytes.

DETAILED DESCRIPTION:
This study aims to test the extent of association of FLIM parameters of cumulus cells with clinical outcomes (clinical pregnancy, ongoing pregnancy at 12 weeks, and live birth) of the embryos that result from the enclosed oocytes.

Participants will be consented to and pre-signed following standard regimens of IVFMD, My Duc Hospital and IVFMD PN, My Duc Phu Nhuan Hospital. The standard is for patients with at least 8 follicles ≥ 10 mm on ultrasonography at the induced ovulation date.

Cumulus samples (CCs) will be collected following the protocol on the day of oocyte pick up (OPU), being assigned with the same number as the oocyte from which it was collected, and vitrified with a Cryotech kit until FLIM measurements are performed.

Insemination will be performed by using ICSI, 3 - 4 hours after oocyte retrieval. A sample of CCs will be sliced off the cumulus mass of each oocyte judged to be mature based on the cumulus mass disposition (absence of tight corona layers). The remaining cumulus cells will be stripped from the OCCs using hyaluronidase. Only mature oocytes will be inseminated.

The fertilization check will be performed under an inverted microscope for a period of 16-18 hours after insemination. On day 3, embryo evaluation will be performed at a fixed time point 66±2 hours after fertilization and, for day 5/6 transfers at 116±2 hours or 140±2 hours, respectively, using the Istanbul consensus. Freeze-all strategy for day 5 embryo will be applied and the first frozen embryo transfer cycle is single embryo transfer.

On the other hand, the investigators will stratify embryos into two groups based on the measured FLIM parameters from their associated cumulus cells, corresponding to the "high" 35% and "low" 65% of metabolic scores.

The investigators aim for embryos in the "high" metabolic scoring group to have a 10% higher live birth rate than controls. Assuming a current live birth rate of 32%, this corresponds to a hoped-for 42% live birth rate in the "high" group (and a 25% live birth rate in the "low" group). A total of 450 patients are required to detect an effect of this size (power 0.90, two-sided alpha 5%).

The primary endpoint of the study will be the live birth rate after the first embryo transfer of the started treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Having any number of IVF/ICSI attempts
* Ovarian stimulation with any stimulation protocol
* Patients with at least 8 follicles ≥ 10 mm on ultrasonography at induced ovulation date
* Agreed to freeze-all day 5-6 embryos
* Agreed to have a single day 5-6 embryo transfer.
* Agreed to participate in the research (signed the consent form)

Exclusion Criteria:

* In vitro maturation (IVM) cycles
* Cycles using testicular biopsy or epididymal sperm
* Cycles not having an oocyte freeze-all cycle
* Cycles using standard insemination
* Participating in another research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Vietnamese infertile women who have IVF/ICSI cycle with at least 8 follicles ≥ 10 mm on ultrasonography at induced ovulation date agreed to freeze-all day 5-6 embryos at IVFMD and IVFMD PN will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate after one frozen embryo transfer cycle | After 24 week's gestation
  The birth of at least one newborn, after 24 week's gestation that exhibits any sign of life, such as respiration, heartbeat, umbilical pulsation, or movement of voluntary muscles

SECONDARY OUTCOMES:
Positive pregnancy test | At 2 weeks after embryo placement
  Positive pregnancy test is defined as a serum human chorionic gonadotropin level greater than 25 mIU/mL after2 weeks after embryo placement of the first transfer
Clinical pregnancy | 7 week's gestation
  The presence of at least one gestational sac on ultrasound at 7 week's gestation with the detection of heartbeat activity, after the completion of the first transfer
Implantation rate | 3 weeks after the first transfer
  Implantation rate is defined as the number of gestational sacs per number of embryos transferred 3 weeks after the first transfer
Ongoing pregnancy | At 10 weeks after embryo placement
  Having at least 1 gestational sac on ultrasound at 12 weeks' gestation with heart beat activity

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, MCE, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Ho Chi Minh City, Vietnam

REFERENCES:
- [Result] Fauser BC. Towards the global coverage of a unified registry of IVF outcomes. Reprod Biomed Online. 2019 Feb;38(2):133-137. doi: 10.1016/j.rbmo.2018.12.001. Epub 2018 Dec 14. No abstract available. PMID 30593441
- [Result] Dumollard R, Duchen M, Carroll J. The role of mitochondrial function in the oocyte and embryo. Curr Top Dev Biol. 2007;77:21-49. doi: 10.1016/S0070-2153(06)77002-8. PMID 17222699
- [Result] May-Panloup P, Boucret L, Chao de la Barca JM, Desquiret-Dumas V, Ferre-L'Hotellier V, Moriniere C, Descamps P, Procaccio V, Reynier P. Ovarian ageing: the role of mitochondria in oocytes and follicles. Hum Reprod Update. 2016 Nov;22(6):725-743. doi: 10.1093/humupd/dmw028. Epub 2016 Aug 25. PMID 27562289
- [Result] Babayev E, Seli E. Oocyte mitochondrial function and reproduction. Curr Opin Obstet Gynecol. 2015 Jun;27(3):175-81. doi: 10.1097/GCO.0000000000000164. PMID 25719756
- [Result] Scott R 3rd, Zhang M, Seli E. Metabolism of the oocyte and the preimplantation embryo: implications for assisted reproduction. Curr Opin Obstet Gynecol. 2018 Jun;30(3):163-170. doi: 10.1097/GCO.0000000000000455. PMID 29708901
- [Result] Chakraborty S, Nian FS, Tsai JW, Karmenyan A, Chiou A. Quantification of the Metabolic State in Cell-Model of Parkinson's Disease by Fluorescence Lifetime Imaging Microscopy. Sci Rep. 2016 Jan 13;6:19145. doi: 10.1038/srep19145. PMID 26758390
- [Result] Becker W. Fluorescence lifetime imaging--techniques and applications. J Microsc. 2012 Aug;247(2):119-36. doi: 10.1111/j.1365-2818.2012.03618.x. Epub 2012 May 24. PMID 22621335
- [Result] Sanchez T, Wang T, Pedro MV, Zhang M, Esencan E, Sakkas D, Needleman D, Seli E. Metabolic imaging with the use of fluorescence lifetime imaging microscopy (FLIM) accurately detects mitochondrial dysfunction in mouse oocytes. Fertil Steril. 2018 Dec;110(7):1387-1397. doi: 10.1016/j.fertnstert.2018.07.022. Epub 2018 Nov 14. PMID 30446247
- [Result] Sanchez T, Zhang M, Needleman D, Seli E. Metabolic imaging via fluorescence lifetime imaging microscopy for egg and embryo assessment. Fertil Steril. 2019 Feb;111(2):212-218. doi: 10.1016/j.fertnstert.2018.12.014. PMID 30691624
- See also: T. H. F. and E. A. (HFEA), "Fertility treatment 2019: trends and figures," 2021. — https://www.hfea.gov.uk/about-us/publications/research-and-data/fertility-treatment-2019-trends-and-figures/